CLINICAL TRIAL: NCT03882177
Title: StAT-TB (Statin Adjunctive Therapy for TB): A Phase 2b Dose-finding Study of Pravastatin in Adults With Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: StAT-TB; 38558 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Tuberculosis; Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary | interventions — Pravastatin; Vitamin B 6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: Pravastatin (40 mg) and Rifafour (Experimental): Participants will receive pravastatin (40 mg) and Rifafour daily for 14 days. Pravastatin will be given alone on Day 1, and pravastatin + Rifafour will be given on Days 2-15.
  Vitamin B6 will be added to each of the regimens.
  Interventions: Drug: Pravastatin; Drug: Rifafour; Dietary Supplement: Vitamin B6
- Arm 2: Pravastatin (80 mg) and Rifafour (Experimental): Participants will receive pravastatin (80 mg) and Rifafour daily for 14 days. Pravastatin will be given alone on Day 1, and pravastatin + Rifafour will be given on Days 2-15.
  Vitamin B6 will be added to each of the regimens.
  Interventions: Drug: Pravastatin; Drug: Rifafour; Dietary Supplement: Vitamin B6
- Arm 3: Pravastatin (120 mg) and Rifafour (Experimental): Participants will receive pravastatin (120 mg) and Rifafour daily for 14 days. Pravastatin will be given alone on Day 1, and pravastatin + Rifafour will be given on Days 2-15.
  Vitamin B6 will be added to each of the regimens.
  (Arm 3 will only be recruited if pravastatin 80 mg is well tolerated and safe, yet drug exposures are significantly reduced due to the known interaction with rifampin.)
  Interventions: Drug: Pravastatin; Drug: Rifafour; Dietary Supplement: Vitamin B6
- Arm 4: Pravastatin (160 mg) and Rifafour (Experimental): Participants will receive pravastatin (160 mg) and Rifafour daily for 14 days. Pravastatin will be given alone on Day 1, and pravastatin + Rifafour will be given on Days 2-15.
  Vitamin B6 will be added to each of the regimens.
  (Arm 4 will only be recruited if pravastatin 120 mg is well tolerated and safe, yet drug exposures are significantly reduced due to the known interaction with rifampin.)
  Interventions: Drug: Pravastatin; Drug: Rifafour; Dietary Supplement: Vitamin B6

INTERVENTIONS:
Drug: Pravastatin — Tablets, administered orally
Drug: Rifafour — Fixed-dose combination (isoniazid, rifampin, pyrazinamide, and ethambutol) tablets, administered orally
Dietary Supplement: Vitamin B6 — Administered orally.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of pravastatin adjunctive therapy when combined with the standard tuberculosis (TB) treatment regimen in adults with TB.

DETAILED DESCRIPTION:
This study will assess the safety, tolerability, and pharmacokinetics of pravastatin adjunctive therapy when combined with the standard TB treatment regimen in adults with drug-sensitive TB. The pharmacokinetic data for pravastatin will be used to choose a dose to be studied as adjunctive TB treatment in subsequent trials.

This study is a dose-escalation trial, and participants will be sequentially enrolled into four study arms. Participants will receive standard anti-TB therapy (Rifafour) and pravastatin daily for 14 days. Pravastatin will be given alone on Day 1, and pravastatin + Rifafour will be given on Days 2-15.

Total study duration for participants will be 30 days, during which time participants will attend several study visits. Study visits may include sputum specimen collection, blood and urine collection, lung function testing, and pharmacokinetic assessments. All study participants will be referred appropriately to continue standard TB treatment at study completion.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Clinical signs and symptoms of pulmonary tuberculosis
* Abnormal chest radiograph consistent with pulmonary tuberculosis
* At least one sputum positive for M. tuberculosis by Xpert MTB/RIF with a cycle threshold (Ct) less than 28.
* Documentation of HIV status
* Weight greater than or equal to 45 kg
* Karnofsky score of at least 60
* Ability to provide informed consent
* Ability to adhere to study follow-up visits
* Negative pregnancy test in women of child-bearing age
* Ability to adhere to contraceptive requirements and willing to use two forms of contraception: 1) a double barrier method to prevent pregnancy (i.e. use of a condom with either diaphragm or cervical cap) or 2) use of an intrauterine device in combination with a barrier contraceptive. The participant must be willing to continue these contraceptive measures throughout the duration of the study and until one week after the last dose of study medication or one week after discontinuation from study medication in case of premature discontinuation.
* Five days or fewer of anti-tuberculosis treatment within the previous 3 months

Exclusion Criteria:

* A history of severe adverse reactions to any statin or any other study agent or contraindications to use of statins.
* Current use of statins or other lipid-lower agents;
* Clinical indication for statin therapy based on cardiovascular risk:

  * Familial hypercholesterolemia
  * Previous history of myocardial infarction or stroke
* For HIV-positive individuals, a CD4+ T-cell count less than 350/mm^3
* Use of antiretroviral drugs
* Hemoglobin concentration less than 8 g/dL;
* Baseline creatinine kinase elevation more than three times the upper limit of normal
* Abnormal baseline laboratory values

  * Baseline alanine aminotransferase (ALT) concentration more than 2.5 times the upper limit of normal (Grade 1)
  * Serum creatinine concentration more than twice the upper limit of normal;
  * Serum total bilirubin level greater than twice the upper limit of normal
  * Platelet count less than 100,000/mm^3
  * Absolute neutrophil count (ANC) less than 1,000/mm^3
* Pregnant or breastfeeding;
* Silico-tuberculosis.
* Currently receiving TB treatment
* Serologies or PCR positive for viral hepatitis (Hepatitis, B, C)
* Concomitant disorders or conditions for which isoniazid, rifampin, pyrazinamide, or ethambutol is contraindicated. These include cirrhosis, acute liver disease of any cause, acute uncontrolled gouty arthritis and peripheral neuropathy.
* Any medical or psychological condition which, in the view of the study investigator, makes study participation inadvisable.
* Infection with an isolate determined to be resistant to rifampin by GeneXpert.
* More than five days of anti-tuberculosis treatment within the previous 3 months
* Planned or current use of cyclosporine, tacrolimus, erythromycin or colchicine
* Central nervous system (CNS) TB
* Extra-pulmonary TB only, not in combination with pulmonary TB
* History of TB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petros C. Karakousis, MD, Principal Investigator — Johns Hopkins University; Richard E. Chaisson, MD, Principal Investigator — Johns Hopkins University; Neil Martinson, MD, MPH, Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- PHRU Non-Network CRS, Johannesburg, Gauteng, South Africa

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Pravastatin (40 mg) and Rifafour: Participants will receive pravastatin (40 mg) and Rifafour daily for 14 days. Pravastatin will be given alone on Day 1, and pravastatin + Rifafour will be given on Days 2-15.
  Vitamin B6 will be added to each of the regimens.
  Pravastatin: Tablets, administered orally
  Rifafour: Fixed-dose combination (isoniazid, rifampin, pyrazinamide, and ethambutol) tablets, administered orally
  Vitamin B6: Administered orally.
- Arm 2: Pravastatin (80 mg) and Rifafour: Participants will receive pravastatin (80 mg) and Rifafour daily for 14 days. Pravastatin will be given alone on Day 1, and pravastatin + Rifafour will be given on Days 2-15.
  Vitamin B6 will be added to each of the regimens.
  Pravastatin: Tablets, administered orally
  Rifafour: Fixed-dose combination (isoniazid, rifampin, pyrazinamide, and ethambutol) tablets, administered orally
  Vitamin B6: Administered orally.
- Arm 3: Pravastatin (120 mg) and Rifafour: Participants will receive pravastatin (120 mg) and Rifafour daily for 14 days. Pravastatin will be given alone on Day 1, and pravastatin + Rifafour will be given on Days 2-15.
  Vitamin B6 will be added to each of the regimens.
  (Arm 3 will only be recruited if pravastatin 80 mg is well tolerated and safe, yet drug exposures are significantly reduced due to the known interaction with rifampin.)
  Pravastatin: Tablets, administered orally
  Rifafour: Fixed-dose combination (isoniazid, rifampin, pyrazinamide, and ethambutol) tablets, administered orally
  Vitamin B6: Administered orally.
- Arm 4: Pravastatin (160 mg) and Rifafour: Participants will receive pravastatin (160 mg) and Rifafour daily for 14 days. Pravastatin will be given alone on Day 1, and pravastatin + Rifafour will be given on Days 2-15.
  Vitamin B6 will be added to each of the regimens.
  (Arm 4 will only be recruited if pravastatin 120 mg is well tolerated and safe, yet drug exposures are significantly reduced due to the known interaction with rifampin.)
  Pravastatin: Tablets, administered orally
  Rifafour: Fixed-dose combination (isoniazid, rifampin, pyrazinamide, and ethambutol) tablets, administered orally
  Vitamin B6: Administered orally.
Period: Overall Study
Arm/Group | Arm 1: Pravastatin (40 mg) and Rifafour | Arm 2: Pravastatin (80 mg) and Rifafour | Arm 3: Pravastatin (120 mg) and Rifafour | Arm 4: Pravastatin (160 mg) and Rifafour
Started | 10 | 6 | 0 | 0
Completed | 10 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled and no data was collected in the 120mg and 160mg pravastatin arms due to early termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Pravastatin (40 mg) and Rifafour | Arm 2: Pravastatin (80 mg) and Rifafour | Arm 3: Pravastatin (120 mg) and Rifafour | Arm 4: Pravastatin (160 mg) and Rifafour | Total
Number analyzed (Participants) | 10 | 6 | 0 | 0 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.70 (5.35) | 26.83 (7.03) |  |  | 26.75 (5.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 |  |  | 5
  Male | 7 | 4 |  |  | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African/Black | 10 | 6 |  |  | 16
  Coloured | 0 | 0 |  |  | 0
  Indian/Asian | 0 | 0 |  |  | 0
  White | 0 | 0 |  |  | 0
  Other | 0 | 0 |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 10 | 6 |  |  | 16
Weight at Baseline (kg) [Count of Participants; unit: Participants]
  45-49 kg | 1 | 0 |  |  | 1
  50-59 kg | 7 | 4 |  |  | 11
  60-69 kg | 2 | 2 |  |  | 4
HIV Status [Count of Participants; unit: Participants]
  Negative | 10 | 6 |  |  | 16
  Positive | 0 | 0 |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Grade 3 or Higher Adverse Events
Description: Graded using the DAIDS table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017
Time Frame: Measured through Day 30
Population: Participants were not enrolled in Arms 3 and 4 due to early termination.
Measure: Number; unit: AEs Grade 3 or Higher
Arm/Group | Arm 1: Pravastatin (40 mg) and Rifafour | Arm 2: Pravastatin (80 mg) and Rifafour | Arm 3: Pravastatin (120 mg) and Rifafour | Arm 4: Pravastatin (160 mg) and Rifafour
Number analyzed (Participants) | 10 | 6 | 0 | 0
AEs Grade 3 or Higher | 8 | 4 |  |

2. Secondary Outcome: Number of Participants Who Permanently Discontinue Assigned Study Regimen for Any Reason
Description: (Other than new recognition of participant ineligibility based on absence of M. tuberculosis growth in baseline sputum cultures, or growth of M. tuberculosis resistant to rifampin by GeneXpert)
Time Frame: Measured through Day 14
Population: Participants were not enrolled in Arms 3 and 4 due to early termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Pravastatin (40 mg) and Rifafour | Arm 2: Pravastatin (80 mg) and Rifafour | Arm 3: Pravastatin (120 mg) and Rifafour | Arm 4: Pravastatin (160 mg) and Rifafour
Number analyzed (Participants) | 10 | 6 | 0 | 0
Participants | 10 | 6 | 0 | 0

ADVERSE EVENTS:
Time Frame: Measured up to 30 days
Description: Adverse Events and Serious Adverse Events graded using the DAIDS table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017
Arm/Group | Arm 1: Pravastatin (40 mg) and Rifafour | Arm 2: Pravastatin (80 mg) and Rifafour | Arm 3: Pravastatin (120 mg) and Rifafour | Arm 4: Pravastatin (160 mg) and Rifafour
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/10 | 1/6 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 5/10 | 3/6 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Pravastatin (40 mg) and Rifafour (N=10) | Arm 2: Pravastatin (80 mg) and Rifafour (N=6) | Arm 3: Pravastatin (120 mg) and Rifafour (N=0) | Arm 4: Pravastatin (160 mg) and Rifafour (N=0)
Elevated Uric Acid (Investigations) | 3 (3) | 1 (1) | NA | NA
Elevated liver enzymes (ALT/AST) (Investigations) | 1 (1) | 0 (0) | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Pravastatin (40 mg) and Rifafour (N=10) | Arm 2: Pravastatin (80 mg) and Rifafour (N=6) | Arm 3: Pravastatin (120 mg) and Rifafour (N=0) | Arm 4: Pravastatin (160 mg) and Rifafour (N=0)
Decreased hemoglobin level (Investigations) | 1 (1) | 0 (0) | NA | NA
Elevated creatinine kinase (Investigations) | 1 (1) | 0 (0) | NA | NA
Elevated liver enzymes (ALT/AST) (Investigations) | 1 (1) | 0 (0) | NA | NA
Elevated uric acid (Investigations) | 2 (2) | 3 (3) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT03882177/Prot_SAP_000.pdf